CLINICAL TRIAL: NCT06241937
Title: A Prospective, Longitudinal Study of a Revised Firearm Safety Curriculum for Pre-Clinical Medical Students
Brief Title: Medical Student Firearm Safety Counseling Follow-Up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Gary Holland, MD, Distinguished Professor of Ophthalmology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-000968A
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Medical Student Knowledge of Firearm Violence Epidemiology; Medical Student Knowledge About Firearm Safety Procedures; Medical Student-initiated Clinical Firearm Safety Counseling
Keywords: Firearm; Firearm Safety Counseling; Suicide Prevention; Medical Education
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Survey responses and student performances during the simulated patient encounter for members of the DGSOM Class of 2027 who consent to study participation will be compared with those of the students in the DGSOM Classes of 2023 and 2024 in the investigators' previous study of firearm safety counseling training, who consented to the future use of their study data (ClinicalTrials.Gov ID: NCT05242627). Surveys and simulated patient encounter scenario will be identical in both studies, to allow for optimal comparison to the historical controls.
Masking Description: The simulated patient encounter used for this study is a regular component of the DGSOM curriculum used to assess student skills in history taking and physical examination. Students will not be told specifically before the activity that one of the assessments will be whether or not they counseled the simulated patient about firearm safety. Following the activity, the students will be invited to provide informed consent for investigators to view video recordings of the activity for educational research. The firearm screening and counseling performance will not be a factor in a student's grade for the simulated patient encounter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DGSOM Class of 2027 (Experimental)
  Interventions: Behavioral: Expanded Clinical Firearm Safety Counseling Training

INTERVENTIONS:
Behavioral: Expanded Clinical Firearm Safety Counseling Training — Members of the DGSOM class of 2027 will participate in a mandatory 3.5 hour training session as a part of the regular curriculum that will include: (1) didactic information on firearm violence epidemiology; (2) suicide epidemiology and introduction to lethal means restriction; (3) firearm safety counseling techniques; (4) a panel of firearm violence survivors / trauma interventionists; and (5) a small group session with discussions of the aforementioned topics and a demonstration of a patient encounter using a standardized patient actor depicting a clinical scenario warranting firearm safety counseling. The training will be taught by faculty members, invited subject matter experts, senior medical students, and the DGSOM Standardized Patient Program.

SUMMARY:
The preclinical curriculum related to firearm violence and safety counseling at the UCLA David Geffen School of Medicine (DGSOM) has been expanded for the Class of 2027, informed by the results and conclusions of an initial study of firearm safety counseling by medical students (ClinicalTrials.gov ID: NCT05242627), which was conducted by the present study team. The 1-hour firearm safety counseling training session used in that study will be taught again to first-year medical students in the Class of 2027, but training will be augmented with additional instruction; the Class will receive additional comprehensive instruction on suicide risk assessment and will participate in small group breakout sessions, to facilitate the opportunity for students to discuss issues related to firearm violence as a public health issue and to practice firearm safety counseling with standardized patient actors (SPs). Assessment of access to firearms and firearm safety counseling will be added as a standard component of the Social History that students are taught to obtain from patients during clinical examinations. The goal of the expanded training is to increase the prevalence of medical student counseling when they are conducting a history and physical examination in a simulated patient encounter with an SP 6 months after the initial training session, when compared to results from the initial study. The scenario provided to the SP will be identical to that used in the initial study and is a situation in which firearm safety counseling is warranted.

Students will participate in a survey to ascertain their knowledge of firearm violence and their attitudes about physician counseling about firearm safety, prior to formal instruction. Informed consent will be obtained from students to use their responses in educational research. Following the didactic and small group sessions, students will be asked to complete a post-training survey that is similar to the original survey, as a means of assessing knowledge gained and any change in attitudes about physician counseling. The simulated patient encounter will occur approximately 6 months later, after which students will complete another survey to determine retention of knowledge and their experience during the simulated patient encounter. Students will not be told before the encounter that they will be evaluated regarding firearm safety counseling. The SP will identify which students did and did not raise the issue of firearm safety. Videos recorded of each students' sessions (routinely obtained for grading purposes) will be viewed by investigators for those students who provide informed consent, to determine the quality of counseling, if it was conducted.

Results from this follow-up study will be compared to the results of the initial study as a historical control, to determine whether augmentation of firearm safety counseling training above a 1-hour didactic session increases firearm safety counseling by medical students in a clinical setting and whether it improves retention of knowledge about firearm violence.

ELIGIBILITY:
Eligibility Criteria is limited to being a member of the DGSOM Class of 2027.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of medical student screening for access to firearms and counselling about firearm safety. | 1 Day
  The proportion of first-year medical students in the Class of 2027 who assess for access to firearms and counsel about firearm safety in a simulated patient encounter will be based on reporting by the simulated patient actor after the activity, for students who consent to use of data from the activity for educational research.
Medical Student Knowledge about Firearm violence and Attitudes about Physician Counseling. | 6 months
  Data will be collected from student surveys conducted prior to training, immediately after training, and 6 months after training, the latter administered immediately following the simulated patient encounter. Students will be invited to provide informed consent for use of survey data for educational research.
Firearm Safety Counseling | 1 Day
  For students who consent to use of data recorded from videos of their simulated patient encounter, investigators will score the quality of the counseling, if performed, based on prospectively defined criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- David Geffen School of Medicine at UCLA, Los Angeles, California, United States